CLINICAL TRIAL: NCT00095745
Title: A Multicenter, Long-Term, Open-label, Study to Assess the Safety and Tolerability of Aripiprazole as an Adjunctive Therapy in the Treatment of Outpatients With Major Depressive Disorder
Brief Title: A Long-Term Study of Aripiprazole in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN138-164
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2011-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Antidepressive Agents; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antidepressant + Aripiprazole (No Intervention)
  Interventions: Drug: Antidepressant + Aripiprazole

INTERVENTIONS:
Drug: Antidepressant + Aripiprazole — Antidepressant Caps/Tablets Aripiprazole Tablets, Oral, 2-30mg Aripiprazole, once daily, 52-weeks.
  Other Names: Abilify

SUMMARY:
This trial is a 52-week safety study to evaluate the safety of adjunctive aripiprazole in outpatients with major depressive disorder who have experienced an incomplete response to an ongoing antidepressant trial.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 years or older
* Experiencing Major Depressive Disorder with a duration of minimally 8 weeks.
* Treatment history of an inadequate response to at least one and no more than four antidepressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2004-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Safety assessments | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (58):
- United States (58):
  - Local Institution, Mesa, Arizona
  - Local Institution, Peoria, Arizona
  - Local Institution, Beverly Hills, California
  - Local Institution, Burbank, California
  - Local Institution, Encino, California
  - Local Institution, Garden Grove, California
  - Local Institution, National City, California
  - Local Institution, Orange, California
  - Local Institution, Pasadena, California
  - Local Institution, Riverside, California
  - Local Institution, San Diego, California
  - Local Institution, Denver, Colorado
  - Local Institution, Farmington, Connecticut
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Gainesville, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Orlando, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Smyrna, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Edwardsville, Illinois
  - Local Institution, Oakbrook Terrace, Illinois
  - Local Institution, Terre Haute, Indiana
  - Local Institution, Overland Park, Kansas
  - Local Institution, Wichita, Kansas
  - Local Institution, Lexington, Kentucky
  - Local Institution, Rockville, Maryland
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Farmington Hills, Michigan
  - Local Institution, Okemos, Michigan
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Brooklyn, New York
  - Local Institution, New York, New York
  - Local Institution, Staten Island, New York
  - Local Institution, Chapel Hill, North Carolina
  - Local Institution, Raleigh, North Carolina
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Toledo, Ohio
  - Local Institution, Portland, Oregon
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, East Providence, Rhode Island
  - Local Institution, Charleston, South Carolina
  - Local Institution, Memphis, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Woodstock, Vermont
  - Local Institution, Arlington, Virginia
  - Local Institution, Charlottesville, Virginia
  - Local Institution, Herndon, Virginia
  - Local Institution, Richmond, Virginia
  - Local Institution, Bellevue, Washington
  - Local Institution, Seattle, Washington
  - Local Institution, Morgantown, West Virginia
  - Local Institution, Brown Deer, Wisconsin
  - Local Institution, Middleton, Wisconsin

REFERENCES:
- [Derived] Clayton AH, Baker RA, Sheehan JJ, Cain ZJ, Forbes RA, Marler SV, Marcus R, Berman RM, Thase ME. Comparison of adjunctive use of aripiprazole with bupropion or selective serotonin reuptake inhibitors/serotonin-norepinephrine reuptake inhibitors: analysis of patients beginning adjunctive treatment in a 52-week, open-label study. BMC Res Notes. 2014 Jul 18;7:459. doi: 10.1186/1756-0500-7-459. PMID 25037144